CLINICAL TRIAL: NCT05411523
Title: A Prospective Observational Study Assessing Efficacy of 10-kHz Spinal Cord Stimulation for the Treatment of Chemotherapy-Induced Peripheral Neuropathy
Brief Title: Assessing Effect of Spinal Cord Stimulation on Pain and Quality of Life With Chemotherapy-Induced Peripheral Neuropathy
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 22-001218; NCI-2022-02976 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Chemotherapy-Induced Peripheral Neuropathy; Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Spinal Cord Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (spinal cord stimulation, questionnaires): Patients receiving spinal cord stimulation therapy complete questionnaires over 30 minutes at baseline and at 3, 6, and 12 months.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Spinal Cord Stimulation

INTERVENTIONS:
Other: Quality-of-Life Assessment — Complete quality of life assessment
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaires
Procedure: Spinal Cord Stimulation — Receive spinal cord stimulation therapy
  Other Names: SCS

SUMMARY:
This study examines how spinal cord stimulation (SCS) affects pain level and quality of life in patients experiencing chemotherapy-induced peripheral neuropathy (CIPN). CIPN is a nerve problem and one of the potential side effects of chemotherapy that causes pain, numbness, tingling, swelling, or muscle weakness in different parts of the body. CIPN usually begins in the hands or feet and gets worse over time. SCS is a type of therapy that has proven to be effective in treating numerous non-malignant pain disorders including failed back surgery syndrome, refractory angina, limb ischemia, complex regional pain syndrome, and diabetic peripheral neuropathy. SCS may also be useful in patients with CIPN. This study evaluates how SCS affects pain and quality of life in patients undergoing spinal cord stimulation for CIPN.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To measure percentage of responders who had at least 50% reduction in lower extremity pain at 6 months.

II. To measure overall improvement in neurological assessment at 6 months. III. To measure secondary metrics including change in perceived global change/satisfaction, health-related quality of life, and sleep disturbance.

IV. To determine if there are any significant adverse events encountered with spinal cord stimulation (SCS) therapy for cancer-related pain.

OUTLINE:

Patients receiving spinal cord stimulation therapy complete questionnaires over 30 minutes at baseline and at 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients greater than or equal to 18 years of age who have been clinically diagnosed with CIPN for greater than six months after stopping chemotherapy
* Average pain intensity >= 5 on 11-point numeric rating scale (NRS) in the lower extremities at enrollment
* Failed conventional medication management with at least two neuropathic pain medications
* Have electrophysiological evidence of length-dependent peripheral neuropathy
* Underwent a 10-kHz spinal cord stimulator trial for a primary indication of CIPN and reported a successful trial of at least 75% reduction in pain intensity
* Have stable neurological status
* Be on a stable analgesic regimen
* Be an appropriate candidate for surgical procedures required in this study
* Be able to read and understand English-written questionnaires and sign an informed consent form in English
* Be willing and capable of giving informed consent
* Be willing and able to complete study-related requirements, procedures, and visits

Exclusion Criteria:

* Patient refusal to be included in study
* Presence of lower limb mononeuropathy
* History of lower limb amputation or ulceration
* Presence of another painful condition that is unrelated to CIPN and that is not intended to be treated in this study
* Body mass index (BMI) >= 40
* Omeprazole (OME) > 120 mg
* Progressive neurological disease (multiple sclerosis, chronic inflammatory demyelinating polyneuropathy, rapidly progressive arachnoiditis, brain or spinal cord tumor, central deafferentation syndrome, complex regional pain syndrome, acute herniating disc, severe spinal stenosis)
* Certain comorbidities: coagulation/bleeding disorders, diminished capacity from cardiac/pulmonary disease
* Obtaining another interventional procedure unrelated to SCS to treat limb pain
* Have ongoing metastatic malignant neoplasm or untreated local malignant neoplasm. Included patients must be deemed as in remission per discretion of treating oncologist
* Have a life expectancy of less than one year
* Have untreated addiction or dependency to medications, alcohol, or illicit drugs
* Have active, disruptive, and/or unstable psychological or psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with CIPN.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | At 6 months
  Percentage of patients who experience >= 50% improvement of pain intensity on numeric rating scale score at 6 months compared to baseline. Paired t-test test will be carried out to compare questionnaire scores between each follow-up time point and baseline. All p-values will be reported as two-sided. Statistical Packages for Social Sciences (SPSS) software will be used for statistical analysis.

SECONDARY OUTCOMES:
Pain intensity | At 3 months and 12 months
  Percentage of patients who experience >= 50% improvement of pain intensity at 3 months and 12 months compared to baseline. Paired t-test test will be carried out to compare questionnaire scores between each follow-up time point and baseline. All p-values will be reported as two-sided. SPSS software will be used for statistical analysis.
Neuropathy assessment | At baseline and 6 months
  Assessed with Modified Toronto Clinical Neuropathic Pain Assessment performed by clinicians via a standardized neurological examination and scale. Paired t-test test will be carried out to compare questionnaire scores between each follow-up time point and baseline. All p-values will be reported as two-sided. SPSS software will be used for statistical analysis.
Neuropathic pain severity | At baseline and 6 months
  Assessed with Neuropathy Pain Scale, a comprehensive questionnaire with 11 items assessing components of neuropathic pain. Paired t-test test will be carried out to compare questionnaire scores between each follow-up time point and baseline. All p-values will be reported as two-sided. SPSS software will be used for statistical analysis.
Perceived change/satisfaction | At baseline and 3, 6, and 12 months
  Patient Global Impression Scale reflects patient satisfaction and patient impression regarding the efficacy of the treatment or intervention. Graded on a 7-point scale. Paired t-test test will be carried out to compare questionnaire scores between each follow-up time point and baseline. All p-values will be reported as two-sided. SPSS software will be used for statistical analysis.
Health-related quality of life | At baseline and 3, 6, and 12 months
  Assessed using the European Quality of Life Five Dimension Five Level Scale Questionnaire, a validated scale that measures domains of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Paired t-test test will be carried out to compare questionnaire scores between each follow-up time point and baseline. All p-values will be reported as two-sided. SPSS software will be used for statistical analysis.
Sleep issues | At baseline and 3, 6, and 12 months
  Assessed using the Medical Outcomes Study sleep scale, a 9-item questionnaire. Higher scores indicate poorer sleep quality. Paired t-test test will be carried out to compare questionnaire scores between each follow-up time point and baseline. All p-values will be reported as two-sided. SPSS software will be used for statistical analysis.
Adverse events | At baseline and 3, 6, and 12 months
  Paired t-test test will be carried out to compare questionnaire scores between each follow-up time point and baseline. All p-values will be reported as two-sided. SPSS software will be used for statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan S. D'Souza, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials